CLINICAL TRIAL: NCT06546748
Title: Mini Crush or Double Kissing Crush Stenting Techniques For Complex Left Main Bifurcation Lesions: The EVOLUTE-CRUSH Left Main Study
Brief Title: Mini Crush or Double Kissing Crush Stenting Techniques For Complex Left Main Bifurcation Lesions
Status: Completed | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Collaborators: Koşuyolu Kartal Heart Training and Research Hospital (Other); Basaksehir Cam & Sakura City Hospital (Unknown); Medipol University (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Bağcılar Training and Research Hospital (Unknown); Ankara Etlik City Hospital (Other Government); Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Guner, Associate Professor of Cardiology, Istanbul Mehmet Akif Ersoy Educational and Training Hospital
Other Study IDs: 2024.04-42
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Left Main Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mini-crush Stenting Group
- Double kissing-crush Stenting Group

SUMMARY:
The Crush technique has evolved significantly since its introduction to the literature by Colombo et al in 2003, with multiple iterations including mini-crush (MC) and double kissing-crush (DKC) stenting techniques. The main principle of crush techniques for complex bifurcation lesions is to protrude the side branch (SB) stent towards the main branch to adequately cover the SB ostium and minimize the risk of SB ostium restenosis. It was noticed that the 4-5 mm protrusion of the SB stent resulted in a large volume of the crushed stent and the technique was modified into MC which aimed for approximately 1-2 mm protrusion by Galassi et al in 2007. Despite all the disadvantages of the crush technique, the final kissing balloon inflation (KBI) rate of this technique, along with several iterations has been up to 98%. Moreover, a recent meta-analysis showed that MC was associated with a reduction in risk of major cardiovascular events compared to provisional stenting, crush, and culotte techniques. The DKC is a planned 2-stent technique introduced by Chen et al. The ultimate innovation of this approach is that it is designed to increase the success rate of the final KBI. Provided recrossing of the crushed stent occurs through the proximal cell: another advantage of the DKC technique is to improve the success of KBI. The DKC significantly reduced major cardiovascular events (MACE) compared to provisional stenting, crush, TAP, and culotte. Until now, no clinical investigation has compared the DKC and MC in patients with complex left main bifurcation lesions. Therefore, this study sought to determine the clinical results of DKC and MC stenting techniques under long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* true complex left main bifurcation lesions
* stenting with double kissing-crush or mini-crush as a 2-stent strategy
* participation in regular clinical follow-up

Exclusion Criteria:

* prior history of coronary artery bypass grafting
* cardiogenic shock
* end-stage liver or kidney disease
* allergy to antiplatelet therapy or contrast media
* inappropriate dual antiplatelet therapy
* critically ill with < 1-year life expectancy
* absence of all medical records
* PCI for ST-segment elevation myocardial infarction or in-stent restenosis
* non-complex bifurcation lesions
* treated with a bare metal stent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This multicenter observational study was retrospectively conducted between January 2014 and January 2024, and patients who underwent percutaneous coronary intervention (PCI) for complex left main coronary bifurcation lesions.
Sampling Method: Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events (MACE) | 12 months
  Cardiac death, clinically-driven target lesion revascularization, target vessel myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmet Güner, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Uzun F, Guner A, Hakgor A, Alizade E, Karatas MB, Alici G, Cizgici AY, Sahin I, Gul I, Pusuroglu H, Karaduman A, Akman C, Atas AE, Deniz MF, Tekin DN, Serin E, Kocaaga M, Yasan M, Avci II, Senoz O, Varim P, Dogan A, Dursun A, Unkun T, Cetin I, Gokalp M, Tanik VO, Aktuk IF, Cakal B, Keskin K, Guner EG, Simsek A, Ekiz MA, Uzel ST, Bulus C, Ciloglu K, Goksu MM, Calik AN, Boztosun B. DK-Crush or Mini-Crush Stenting for Complex Left Main Bifurcation Lesions: The Multicenter EVOLUTE-CRUSH LM Registry. J Am Heart Assoc. 2025 Jun 17;14(12):e040166. doi: 10.1161/JAHA.124.040166. Epub 2025 May 21. PMID 40396672